CLINICAL TRIAL: NCT06756867
Title: The Effect of Hand Massage with Violet Oil on Pruritus Level and Quality of Life in Patients
Brief Title: The Effect of Hand Massage with Violet Oil on Pruritus Level and Quality of Life in Patients Receiving Hemodialysis Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, KEVSER ÇAĞLA GURLAŞ, lecturer, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ErciyessaglıkU
Record Dates: First submitted 2024-12-19; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Aromatherapy in Hemodialysis Patients with Itching
Keywords: Quality of Life; hemodialysis; Hand Massage; Pruritus; Violet Oil; Nursing
MeSH Terms: conditions — Pruritus | interventions — fat red 7B; jojoba wax

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Who Masked: Investigator
Masking Description: In the study, pre-test and post-test applications to the sample group will be completed by scholarship students independent of the researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hand massage with violet oil (Experimental): Hand massage with violet oil during hemodialysis session 3 times a week for 6 weeks
  Interventions: Other: hand massage with violet oil
- hand massage with placebo jojoba oil (Placebo Comparator): Hand massage with jojoba oil during hemodialysis session 3 times a week for 6 weeks
  Interventions: Other: hand massage with jojoba oil
- control group (No Intervention): There will be no intervention

INTERVENTIONS:
Other: hand massage with violet oil — In this study, individuals receiving hemodialysis treatment will be massaged with 2% violet oil for 5-7 minutes on the hand on the non-fistula arm during the dialysis session, 3 times a week for six weeks.
  Arms: hand massage with violet oil
Other: hand massage with jojoba oil — Hand massage with jojoba oil for hemodialysis patients 3 times a week for 6 weeks
  Arms: hand massage with placebo jojoba oil

SUMMARY:
Itching is among the common problems in individuals receiving hemodialysis (HD) treatment. Research on the effects of aromatherapy on the symptoms seen in dialysis patients is increasing. Studies in the literature have found findings that aromatherapy reduces skin dryness and itching. This study was an experimental study with randomized intervention, placebo and control groups to determine the effect of a 7-minute massage with 2% violet oil on the hand on the non-fistula arm during the dialysis session, 3 times a week for six weeks, on the level of itching and quality of life in individuals receiving HD treatment. It was planned as. The project will be determined on individuals who are treated in 7 hemodialysis centers in a provincial center and whose itch severity scores are 3 or higher and who meet the inclusion criteria for the study.According to the results, patients who meet the inclusion criteria will be randomly assigned to intervention, placebo and control groups. Considering similar studies in the literature, the number of patients to be sampled was determined as 81 people in total, 27 per group, using the G Power program, provided that alpha = 0.05, power = 0.95 and effect size was 0.8165. Taking into account possible losses, randomization of at least 30 patients will be made to each group. Ethics committee approval and institutional permissions were obtained for the project. Verbal and written informed consent forms will be obtained from individuals. The data of the research will be collected between July 2024 and September 2024. If the required number of samples cannot be reached, the data collection process will be extended. In the study, data will be collected using the patient introduction form, 5 D Itch Scale, Kidney Disease Quality of Life Scale (KDQOLTM-36) and patient follow-up charts. In line with the massage application protocol, in addition to the treatment of patients with high itching scores, hand massage will be applied with violet oil to the individuals in the intervention group and jojoba oil to the placebo group.No action will be taken on the control group. IBM SPSS 24.0 Statistics and Turcosa programs will be used to evaluate the data. Power analysis effect size calculations will be made in the Turcosa program. It is planned to use descriptive (mean, percentage and standard deviation) and analytical statistics (Kolmogorov-Smirnov test, Kruskal-Wallis test, Wilcoxon signed rank test, Mann-Whitney Utest) in data analysis. In comparisons, a p value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 and over,
* willing to participate in the study
* Receiving HD treatment in HD units for at least 6 months and 3 sessions per week,
* Continuing dialysis treatment in the same institution,
* Patients who do not develop allergic reactions such as skin irritation, redness, burning and itching after 30 minutes by applying two drops of the oils used in the study to the outer part of the arm.
* There was no change in the treatment program during the study period,
* Having an itch score of 3 or above on the 5-D Itch Scale,
* Individuals who can understand and communicate with Turkish will be included in the research.

Exclusion Criteria:

* Those who have any disease of the respiratory system,
* Those who have any allergies to the essential oils to be used,
* Having a skin lesion in the area to be massaged,
* Patients who use other TIT methods during the treatment process will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
5D Itch Scale score | 6 weeks
  Elman et al. It was developed by in 2010. The scale evaluates the duration, degree, course, distribution and problems caused by itching experienced in the last two weeks. The total score of the scale varies between the lowest score of 5 (no itching) and the highest score of 25 points (severe itching). Duration, degree, direction and disability of itching are scored between 1 and 5 points.

SECONDARY OUTCOMES:
Kidney Disease Quality of Life Short Form- KDQOLTM-36 | 6 weeks
  It was developed by Hays et al. in 1994 to evaluate the quality of life of individuals receiving dialysis treatment. The original form of the scale consists of 134 items. The scale was shortened to 36 items by the Kidney Disease Quality of Life Improvement Center.The KDQOLTM-36 scale, which evaluates the last month of patients, has 36 items consisting of 5 subscales. SF-12 physical dimension (questions 1,2,3,4,5 and 8), SF-12 mental dimension (questions 6,7,9,10,11 and 12), burden of kidney disease (questions 13-16). It consists of five subscales: questions), symptom list (questions 17-28), and the impact of kidney disease on daily life (questions 29-36). The Likert method was used when scoring each item in the scale. Scores on each dimension range from 0 to 100, with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided